CLINICAL TRIAL: NCT06779565
Title: Comparative Evaluation of Postoperative Pain After Root Canal Preparation With Rotary (Hyflex EDM) vs Reciprocating (Reciproc VDW) System in Molar Teeth: A Randomized Controlled Trial
Brief Title: Comparison of Postoperative Pain After Root Canal Treatment With Rotary vs Reciprocating Systems
Acronym: Post op pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Ahmed Abdullah, Principal investigator, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21MDC
Record Dates: First submitted 2025-01-13; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Comparison of postoperative pain in two groups of patients, who underwent root canal treatment with two different file systems. total 80 patients divided into two groups and given different interventional treatment to monitor pain after treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients did not know which file system was used in their treatment. The investigator also did not disclose the intervention's name; rather, a code name was given to them. The outcomes accessor also did not know the exact name but was provided with a code name.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyflex Group (Active Comparator): These patients underwent root canal treatment due to pain in their molar teeth. The file system used in this arm was Hyflex EDM (Coltene), a rotary file system that moves in a complete 360° rotation and prepares a root canal.
  Interventions: Device: Hyflex EDM system
- Recriproc Group (Active Comparator): These patients underwent root canal treatment due to pain in their molar teeth. The file system used in this arm was Reciproc (VDW), a reciprocating file system that moves in 130° anticlockwise and 50° clockwise motion and prepares a root canal.
  Interventions: Device: Reciproc VDW system

INTERVENTIONS:
Device: Hyflex EDM system — A rotary file system
  Arms: Hyflex Group
Device: Reciproc VDW system — A reciprocating file system
  Arms: Recriproc Group

SUMMARY:
To compare the postoperative pain in patients undergoing root canal instrumentation with two different file systems, Hyflex EDM and Reciproc VDW.

DETAILED DESCRIPTION:
Endodontic postoperative pain is experienced after the procedure of the root canal. It is defined as an unpleasant sensation, of varying degrees, experienced by the patients. Depending upon the individual and other variable, the range of postoperative pain lies between 3% to 58%. Endodontic postoperative pain could occur due to various factors that can be microbial, injured pulp, chemical, or mechanical. Factors that influence pain following a root canal include the presence of preoperative pain, apical debris extrusion, intracanal interappointment dressing extrusion, presence of periapical pathosis, hyper occlusion, and irrigant extrusion.

Although apically extruded debris can be reduced through various means, it cannot be completely avoided. Thus, increasing the incidence of postoperative pain in patients. The debris produced during apical extrusion contains necrotic tissue, dental chips, microbes, pulp tissue, and canal irrigants. The infected debris may disturb the balance between the microbes and the immune system, leading to acute exacerbation.

Manual steel K files tend to produce more debris, causing a high risk of postoperative discomfort. Nickel-titanium rotary instruments powered by the engine have various advantages including; time-saving, preservation of root canal anatomy, and homogeneous preparation of the root canal shape. The debris produced by these instruments is potentially lesser than the manual files. Mainly because they have rotary action and excavate the debris with the help of their flutes. Repeated irrigation along with the action of an engine-driven instrument, has the potential to decrease postoperative pain. Reciproc VDW reciprocating file instruments have potential advantages including reduced fatigue, resistance to fracture, less debris extrusion, good shaping ability, no cross-contamination (single use), and reduced cost.

No previous study has established a relationship between debris extrusion and postoperative care. This study aims to compare the use of the Hyflex EDM and Reciproc VDW systems for preparing permanent human teeth during root canal procedures and their effect on postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unremarkable/ noncontributory medical history
2. Healthy persons between the ages of 18 and 60 years
3. Maxillary and mandibular molar teeth diagnosed with symptomatic irreversible pulpitis.
4. Patients not having taken any medication for 6 hours before treatment
5. No allergies to the drugs or dental material being used in the treatment

Exclusion Criteria:

1. Patients who had taken analgesics on anti-inflammatory drugs within the last 12 hours
2. Pregnant women and patients with immunocompromised health state
3. Patients having severe malocclusion associated with traumatic occlusion
4. Teeth with calcified canals
5. Teeth with periapical radiolucency
6. Teeth with root resorption
7. Teeth previously undergone root canal treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Post Operative Pain | 6 hours - 72 hours
  Document and compare post-operative pain after root canal treatment, after using two different motorized file systems with different mechanisms. The Visual Analog scale (VAS) would be used to assess the pain. The patients would be guided in detail about the VAS scoring system and mark pain according to the readings on VAS. The scale is numbered from 1 - 10, with 1 indicating no pain and 10 indicating worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- 21 MDC, Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: No